CLINICAL TRIAL: NCT04371679
Title: Changes in Cardiac and Pulmonary Hemodynamics as Predictor of Outcome in Hospitalized COVID-19 Patients
Acronym: COVID-HO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, Head of Cardiology, Hasselt University
Other Study IDs: Covid-HO
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endotracheal intubation and ventilation: Patients admitted at ICU that are intubated and ventilated
  Interventions: Other: No interventions planned
- Non-Invasive Ventilation: Patients admitted at ICU who are non-invasively ventilated
  Interventions: Other: No interventions planned

INTERVENTIONS:
Other: No interventions planned — No interventions planned. Observational.

SUMMARY:
The primary objective of the study is to evaluate cardiac and pulmonary hemodynamic changes over time as predictor of disease progression and outcome in COVID-19 patients admitted to ICU.

The primary endpoint is the occurrence of a major event predefined as either: death (all-cause mortality) or discharge from ICU (limit of 4 months).

This is a uni-center prospective observational cohort study with an inclusion period of 2 months. The end of the study is foreseen in 6 months.

DETAILED DESCRIPTION:
Background COVID-19 can lead to a bilateral pneumonia overwhelming the lungs causing dyspnea and respiratory distress. Up to 20% of the infected population is hospitalized and 5% is submitted to the intensive care unit (ICU). Up to 31% of patients in ICU develop sepsis and 61% develop ARDS with a deadly outcome at ICU of 38%. While sepsis typically causes diffuse vasodilation, the pulmonary vasculature resistance in ARDS is high. Although heart failure is per definition not the cause of ARDS, the resulting elevated pressures in the pulmonary circulation affect right and left heart function. Early detection in alterations of cardiac and pulmonary hemodynamics might prompt to actions to prevent ARDS.

Primary objective To evaluate cardiac and pulmonary hemodynamic changes over time as predictor of disease progression and outcome in COVID-19 patients admitted to ICU.

Secondary objective

* Analysis of prognostic factors based on the data at initial presentation
* Performing a trajectory analysis of the time course during ICU stay to determine what leads to optimal outcome - gain insight in the pathophysiology of the cardio-pulmonary evolution of COVID-19 pts
* Feasibility study for the creation of an individualized expected data-trajectory for new cases and continuously updating its visualization in relation to the expected trajectory related to an improved outcome
* Evaluate how Machine Learning, based on manifold learning for quantifying information similarity and its temporal evolution, is able to predict outcome using rich data in a limited number of patients Primary Endpoint

Occurrence of a major event predefined as either:

* Death (all-cause mortality)
* Discharge from ICU (limit of 4 months) Secondary Endpoint
* Decrease of left ventricular (LV) function defined by LV global longitudinal strain (GLS) > 5% (absolute value) and LV S' as compared to the initial evaluation
* Evolution of LV diastolic function related to prognosis - Doppler Data and ML interpretation
* Decrease of right ventricular (RV) function by RV GLS > 5% (absolute values) or decrease of RV S' to an absolute value <9.5 cm/s
* Dynamic RV response to PEEP maneuver to differentiate intrinsic RV dysfunction from excessive PEEP.
* Changes in pulmonary arterial compliance from RVOT-VTI and PASP Methods Uni-center cohort study (Prospective Observational) Duration of the study Duration of the inclusion period: 2 months Duration of participation for each patient: average 4 weeks until death or discharge from ICU Duration of data processing and reports: 4 months Total duration of the study: 6 months

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to ICU that is COVID-19 positive based on rt-PCR
* Ventilated or not ventilated
* No restrictions on age
* No restrictions on comorbidities or a diversity of underlying pathology (malignancies, COPD, …)

Exclusion Criteria:

* Patients that are not COVID-19 tested (rt-PCR) or where the diagnosis is pending.
* Patients that refuse their participation in the study.
* Patients under legal protection, or deprived of their liberty.
* Patients that are so critically ill that a minimum of 1 follow-up is very unlikely to be realised

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive COVID-19 positive patients that are admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Death (all-cause mortality) or discharge from ICU (limit of 4 months) | 4 months
  Covid-19 pneumonia that requires ICU admission can go either way.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Herbots, MD, PhD, Principal Investigator — Hartcentrum Hasselt
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No